CLINICAL TRIAL: NCT01463293
Title: Effects of 4-week Bifidobacterium Lactis HN019 Supplementation on Whole Gut Transit Time and Gastrointestinal Symptoms in Adults With Constipation: A Double-blind, Randomized, Placebo-controlled Dose-ranging Trial
Brief Title: B. Lactis HN019 for Functional Constipation
Acronym: CTT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fonterra Research Centre (Industry)
Collaborators: DuPont Nutrition and Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-SUS-02-FON-02
Record Dates: First submitted 2011-10-28; First posted 2011-11-01 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-06

CONDITIONS: Constipation
Keywords: constipation; probiotic; functional constipation; IBS-C
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-dose probiotic (Experimental): Capsule containing 10 billion cfu B. lactis HN019
  Interventions: Dietary Supplement: B. lactis HN019
- Low dose probiotic (Experimental): Capsule containing 1 billion cfu B. lactis HN019
  Interventions: Dietary Supplement: B. lactis HN019
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: B. lactis HN019 — Capsule containing 10 billion cfu B. lactis HN019 once a day
  Arms: High-dose probiotic
Dietary Supplement: B. lactis HN019 — Capsule containing 1 billion cfu B. lactis HN019 once a day
  Arms: Low dose probiotic
Dietary Supplement: Placebo — Capsule containing no probiotic once a day
  Arms: Placebo

SUMMARY:
This study will investigate the effects of 4-week probiotic supplementation on whole gut transit time and gastrointestinal symptoms in adults with functional constipation.

DETAILED DESCRIPTION:
This prospective, double-blind, randomized, placebo-controlled clinical trial will investigate the effects of 4-week B. lactis HN019 supplementation on whole gut transit time and gastrointestinal symptoms in adults with functional constipation. Participants who meet all study entry criteria will enter a 2-week run-in period. Following successful completion of the run-in period, subjects will be randomized to 4-week supplementation with B. lactis HN019 (10 billion cfu), B. lactis HN019 (1 billion cfu), or placebo. The primary outcome of whole gut transit time will be evaluated with abdominal x-rays on days 0 and 28. Secondary outcomes include IBS-specific questionnaires (administered on days 0 and 28); abdominal pain severity, bowel movement frequency, stool consistency, and adverse events (evaluated daily throughout the study); and overall product satisfaction (evaluated at day 28). Physical activity questionnaires and 24-hour food recalls will be completed periodically during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Body mass index between 18.5 and 34.9 kg/m2
* Self-reported unsatisfactory defecation due to infrequent stools and/or difficult stool passage, which includes at least one of the following: symptoms of straining, difficulty expelling stool, a sense of incomplete evacuation, hard or lumpy stools, prolonged time to stool, or a need for manual maneuvers to pass stool.
* Estimated stool consistency < 4.0 on BSSF (self-reported at screening) within the past month prior to enrollment.
* Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects
* Consent to the study and willing to comply with study product and methods

Exclusion Criteria:

* Major gastrointestinal complication (e.g. Crohn's disease, ulcer)
* Prior abdominal surgery that, in the opinion of the investigator, may present a risk for the subject or confound study results
* Clinically significant underlying systemic illness that may preclude the subject's ability to complete the trial or that may confound the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness)
* Daily consumption of probiotics, prebiotics, fermented milk, and/or yogurt within 2 weeks of screening and throughout the trial other than the provided study products
* Non-laxative constipation medication use within 2 weeks of screening, laxative use within 48 hours of screening (rescue medication allowed for intolerable symptoms during study)
* Daily use of anticholinergic agents, opioid analgesics, calcium supplements, calcium-channel blockers, and NSAIDs
* Anticipated major dietary or exercise changes during the study
* Systemic steroid use
* Eating disorder
* Contraindication to dairy products (e.g., intolerance to lactose or any substance in the study product)
* History of alcohol, drug, or medication abuse
* Pregnant or lactating female, or pregnancy planned during study period
* Participation in another study with any investigational product within 30 days of screening
* Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hardi, MD, Principal Investigator — Capital Digestive Care, LLC
Locations (12):
- United States (12):
  - Arrowhead Family Health Center, Glendale, Arizona
  - Diagnamics, Inc., Encinitas, California
  - Digestive & Liver Disease Specialists, Garden Grove, California
  - StayWell Research, Northridge, California
  - Sprim ALS, San Francisco, California
  - Westlake Medical Research, Westlake Village, California
  - Research Across America, Carrollton, Texas
  - Research Across America, Dallas, Texas
  - Discovery Clinical Trials South Main, Houston, Texas
  - Research Across America, Katy, Texas
  - Village Health Partners, Plano, Texas
  - North Texas Family Medicine, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-dose Probiotic | Low Dose Probiotic | Placebo
Started | 74 | 79 | 71
Completed | 68 | 63 | 59
Not Completed | 6 | 16 | 12
Not completed — Lost to Follow-up | 1 | 4 | 5
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Withdrawal by Subject | 4 | 10 | 5
Not completed — Other | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose Probiotic | Low Dose Probiotic | Placebo | Total
Number analyzed (Participants) | 74 | 79 | 71 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (12.1) | 42.9 (12.0) | 41.1 (12.6) | 41.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 51 | 161
  Male | 18 | 25 | 20 | 63
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian, non-Hispanic | 27 | 35 | 26 | 88
  Asian | 4 | 2 | 6 | 12
  Hispanic | 17 | 11 | 11 | 39
  Native American | 1 | 1 | 0 | 2
  African-American, Black | 19 | 25 | 24 | 68
  Other | 6 | 5 | 4 | 15
Region of Enrollment [Number; unit: participants]
  United States | 74 | 79 | 71 | 224
Height, M [Mean (Standard Deviation); unit: M] | 1.66 (0.12) | 1.68 (0.09) | 1.68 (0.10) | 1.68 (0.10)
Weight, Kg [Mean (Standard Deviation); unit: Kg] | 74.9 (15.2) | 77.5 (15.9) | 74.3 (14.9) | 75.6 (15.0)
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 27.0 (4.2) | 27.4 (4.4) | 26.6 (4.7) | 27.0 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Whole Gut Transit Time
Description: The primary endpoint of this clinical trial is whole gut transit time, which will be assessed using abdominal x-rays on days 0 and 28
Time Frame: 4 weeks
Population: Only 39 out of the 224 enrolled subjects consumed the radio-opaque markers in line with the protocol. Because of the substantial number of protocol deviations and the lack of sufficient evaluable subjects, no further analyses of the study data were performed. The study appears not to have yielded evaluable data.
Arm/Group | High-dose Probiotic | Low Dose Probiotic | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Patient Assessment of Constipation Symptoms (PAC-SYM)
Description: The PAC-SYM tool asks 12 questions on the symptoms of constipation. Subjects will complete the PAC-SYM at days 0 and 28.
Time Frame: 4 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Patient Assessment of Constipation QoL (PAC-QoL)
Description: The PAC-QoL is a 28-question survey that asks questions on their quality of life.
Time Frame: 4 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Bowel Function Index
Description: The Bowel Function Index is a 3-question tool that asks subjects if they have experienced adequate relief of constipation symptoms over the past week. The Bowel Function Index will be completed at days 0 and 28.
Time Frame: 4 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Adequate Relief of Constipation (Yes/no)
Description: Adequate relief of constipation (yes/no) This (yes/no) questionnaire will be completed at days 0 and 28.
Time Frame: 4 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Bowel Movement Frequency
Description: Subjects will record the number of defecations per day in a diary.
Time Frame: 4 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Stool Consistency
Description: Stool consistency will be rated each day in a diary by using the Bristol Stool Scale Form
Time Frame: 4 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Overall Product Satisfaction
Description: At the end of the supplementation period, subjects will be asked to rate their overall satisfaction with the study product's ability to relieve their constipation symptoms on a 5-point ordinal scale
Time Frame: 4 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Adverse Event Frequency
Description: All adverse events, regardless of relationship with investigational product, will be reported during the 4-week follow-up period.
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | High-dose Probiotic | Low Dose Probiotic | Placebo
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/79 | 0/71
Other Adverse Events (participants affected / at risk) | 17/74 | 16/79 | 20/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Probiotic (N=74) | Low Dose Probiotic (N=79) | Placebo (N=71)
Gastrointestinal discomfort (Gastrointestinal disorders) | 3 | 4 | 5
Respriatory symptoms (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1 — Upper respiratory tract infection, common cold, bronchitis
Headache (General disorders) | 1 | 4 | 3
Injury (General disorders) | 1 | 0 | 3
Other (General disorders) | 7 | 6 | 8

LIMITATIONS AND CAVEATS:
A substantial number of protocol violations occurred for the primary end-point. Only 39 out of 224 subjects consumed sufficent radio-opaque markers for baseline and post-intervention transit time.Therefore, the study failed to yield evaluable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less